CLINICAL TRIAL: NCT03097159
Title: Comparison of Costoclavicular Brachial Plexus Block and Supraclavicular Brachial Plexus Block
Acronym: BPB
Status: Withdrawn | Type: Observational
Why Stopped: Surgeon refuse the proposal, so we can's enroll the patients
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Other Study IDs: 106421
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Phrenic Nerve Paralysis
Keywords: costoclavicular block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Costoclavicular block: For anesthesia, this group of patients will be received ultrasound guided costoclavicular block
  Interventions: Procedure: Costoclavicular block
- Supraclavicular block: For anesthesia, this group of patients will be received ultrasound guided supraclavicular block

INTERVENTIONS:
Procedure: Costoclavicular block — Group C for costoclavicular block Group S for supraclavicular block
  Groups: Costoclavicular block

SUMMARY:
The investigator will compare Costoclavicular approach of infraclavicular block and supraclavicular block. Especially, the incidence of phrenic nerve palsy and the quality of block.

DETAILED DESCRIPTION:
Costoclavicular brachial plexus block is a recently developed approach of infraclavicular brachial plexus block. Using ultrasound, all of 3 cords are well visible in single plane. Compared to conventional infraclavicular block, it needs smaller amount of local anesthetics.

Supraclavicular brachial plexus block is known as spinal anesthesia of upper extremities. It provides fast and good quality of anesthesia and analgesia. But some studies showed that there are over 50% of phrenic nerve palsy in supraclavicular block.

In this study, the investigator will compare phrenic nerve palsy incidence and block quality between Costoclavicular block and supraclavicular block using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Scheduled for surgery of hand or forearm

Exclusion Criteria:

* Patient refusal
* Neuromuscular disease
* Pregnancy
* Previous history of surgery of periclavicular region
* Nerve injury history
* Bleeding tendency
* Allergy to local anesthetics
* Other contraindication of regional anesthesia

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery of hand or forearm
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Diaphragm palsy | 30 min
  Using M-mode of ultrasound, compare diaphragm movement pre-block and 30min after block Paralysis : reduced movement more than 75% or paradoxical movement on sniffing Paresis : 25~75% movement Normal : reduced less than 25%

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No